CLINICAL TRIAL: NCT02882438
Title: Glucosamine Sulphate and Ginkgo Biloba for Treating Tinea Pedis
Brief Title: Glucosamine Sulphate and Ginkgo Biloba as Antifungal Activity for Treating Tinea Pedis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahmed A. H. Abdellatif (Other)
Responsible Party: Sponsor-Investigator, Ahmed A. H. Abdellatif, phD and Lectrurer, Pharmaceutics and Industrial Pharmacy, Faculty of Pharmacy, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AlAzharGGATP
Record Dates: First submitted 2015-11-26; First posted 2016-08-29 (Estimated); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Foot Infection Tinea Pedis
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infected group (Active Comparator): A group of volunteers infected with Tinea pedis, Capitis and Versicolor received Ginkgo Biloba in different dosage forms.
  Interventions: Drug: infected group
- Control group (Placebo Comparator): A group of volunteers infected with Tinea pedis, Capitis and Versicolor received placebo without Ginkgo Biloba.
  Interventions: Drug: control group

INTERVENTIONS:
Drug: infected group — Ginkgo Biloba in different dosage forms
  Other Names: Body Spray
  Arms: Infected group
Drug: control group — placebo without Ginkgo Biloba
  Other Names: placebo
  Arms: Control group

SUMMARY:
Tinea Pedis infected the feet of about 20-25% of the world population. Tinea Pedis is a fungal infection of the feet and it is easily spread. Oral therapy is usually used for chronic conditions or when topical treatment has failed. The aim of this study is to prove the antifungal and antibacterial activity of Ginko Biloba (GKB) & Glucosamine (GL) as separate material or both in combination.

DETAILED DESCRIPTION:
Ginko Biloba (GKB) & Glucosamine (GL) were formulated in different dosage forms such as capsules, hydrogel and spray. GKB&GL were in filled in hard gelatin capsules as three formulae (GKB caps, GL caps and both as mixture in caps). Also, GKB&GL were formulated in hydrogel using 2% carbopol 934 as three formulae (GKB only, GL only and both as mixture). The same also were formulated as spray using alcohol, water and glycerol in concentration of 60%, 20% and 20% respectively. The study included 5 trials, involving 35 participants. The oral formulae were tried on 30 participants having Tenia Pedis. Fluconazole was as standard antifungal drug.The antifungal activity of all gel formulae was determined by Agar well-diffusion method. It is also important to follow up and collect data, preferably for six months for local and systemic activity, to establish whether or not the infection recurred or not. In future clinical trials, research should consider the costs of the different treatment approaches.

ELIGIBILITY:
Inclusion Criteria:

* It is important to follow up and collect data, preferably for six months for local and systemic activity of Ginkgo Biloba and Glucosamine, to establish whether the infection recurrent or not.

Exclusion Criteria:

* Larger numbers of participants having different kind of fungal infection are needed to test efficiency drug in order to produce more reliable data.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-09 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Assessment the antifungal activity of Ginkgo Biloba & Glucosamine | six months
  Ginkgo Biloba and Glucosamine will be applied with infected patients even systemically or topically. The results will be compared with control groups to prove the Antifungal Activity.

SECONDARY OUTCOMES:
Stability test for different dosage forms | three months
  Stability test will be studied for dosage forms. The test will carried out by standing the products on shelf life for three months. The stability test will be recorded using high performance liquid chromatography each thee days.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Clinic, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tauber A, Muller-Goymann CC. In vitro model of infected stratum corneum for the efficacy evaluation of poloxamer 407-based formulations of ciclopirox olamine against Trichophyton rubrum as well as differential scanning calorimetry and stability studies. Int J Pharm. 2015 Oct 15;494(1):304-11. doi: 10.1016/j.ijpharm.2015.08.023. Epub 2015 Aug 11. PMID 26276254